CLINICAL TRIAL: NCT01126255
Title: Efficacy of a Topic Therapy With Progesterone Compared to the Conventional Therapy With Clobetasol Propionate in Patients With Vulvar Lichen Sclerosus. A Double Blind, Randomized Phase II Pilot Study.
Brief Title: Progesterone vs Clobetasol Propionate in Vulvar Lichen Sclerosus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment problems
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: PD Dr. med. A. Guenthert, Dep. of Obstetrics and Gynecology, Bern University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 213/08
Record Dates: First submitted 2010-05-07; First posted 2010-05-19 (Estimated); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Vulvar Lichen Sclerosus
Keywords: vulvar lichen sclerosus; progesterone; clobetasol; randomized controlled trial
MeSH Terms: conditions — Vulvar Lichen Sclerosus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Clobetasol propionate 0.05%, topical application, once daily about 2 g, during 12 weeks
  Interventions: Drug: Clobetasol propionate 0.05%
- 2 (Experimental): Progesterone 8%, topical application, once daily about 2 g, during 12 weeks
  Interventions: Drug: Progesterone 8%

INTERVENTIONS:
Drug: Clobetasol propionate 0.05% — Topical application, once daily about 2 g, during 12 weeks
  Arms: 1
Drug: Progesterone 8% — Topical application, once daily about 2 g, during 12 weeks
  Arms: 2

SUMMARY:
This is a randomized trial comparing progesterone with conventional clobetasol propionate in patients with vulvar lichen sclerosus.

DETAILED DESCRIPTION:
Background

A total of 62 female patients with first diagnosis of lichen sclerosus will be treated daily with either topical progesterone 8% or clobetasol propionate 0.05% for 12 weeks. Response to the treatment will be evaluated by macroscopic description of the dermatologic phenotype by using a specific lichen sclerosus score and photography-documentation. The symptoms and quality of life of the patients will be evaluated by standardized questionnaires. Additionally, tissue samples will be taken before and again after 12 weeks of treatment to evaluate the response status.

Objective

The purpose of this study is to compare progesterone with conventional clobetasol propionate in a superiority trial.

Methods

Prospective, randomized, controlled, superiority phase II pilot trial. Patients will be randomized 1:1 to either progesterone or clobetasol propionate, with patients, physicians, assessors and analysts being blinded.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Consent to biopsy at start and end of therapy
* Suspicion of Lichen sclerosus
* Pre-menopausal
* Age ≥18 years

Exclusion Criteria

* Prior surgery at the vulva, with exception of episiotomy
* Pregnancy
* Signs of infection with human papilloma virus at the vulva
* Vulvar intraepithelial neoplasia (VIN)
* Known generalised autoimmune disease
* Lichen sclerosus since childhood
* Prior therapy with topic clobetasol propionate or other immunosuppressives (tacrolimus or pimecrolimus) at the vulva
* Atopic diathesis and/or contact allergy
* Systemic immunosuppressive therapy
* Genital infection within the last four weeks (eg., condyloma acuminata, candidiasis)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Score of the characteristics of Lichen sclerosus based on vulvar efflorescences | at 12 weeks
  The severity of the Lichen sclerosus will be assessed by a metric score, which is based on 6 items (abrasion, hyperkeratosis, rhagades, synechia, sclerosis, atrophy of labia/clitoris) consisting of three levels (0=no signs, 1=few signs, 2=pronounced signs).

SECONDARY OUTCOMES:
Patient-reported symptoms | at baseline
  The patient will report the following symptoms on a scale from 0 to 10 pruritus, burning or pain, sore.
Quality of life | at baseline
  The patient will report quality of life on the SF12 questionnaire.
Adverse events | at baseline
  The tolerability of the topical treatment will be assessed by all adverse events occuring at the site of application.
Patient-reported symptoms | at 6 weeks
  The patient will report the following symptoms on a scale from 0 to 10: pruritus, burning or pain, sore.
Patient-reported symptoms | at 12 weeks
  The patient will report the following symptoms on a scale from 0 to 10: pruritus, burning or pain, sore.
Patient-reported symptoms | at 18 weeks
  The patient will report the following symptoms on a scale from 0 to 10 pruritus, burning or pain, sore.
Patient-reported symptoms | at 24 weeks
  The patient will report the following symptoms on a scale from 0 to 10 pruritus, burning or pain, sore.
Quality of life | at 12 weeks
  The patient will report quality of life on the SF12 questionnaire.
Quality of life | at 24 weeks
  The patient will report quality of life on the SF12 questionnaire.
Adverse events | at 6 weeks
  The tolerability of the topical treatment will be assessed by all adverse events occuring at the site of application.
Adverse events | at 12 weeks
  The tolerability of the topical treatment will be assessed by all adverse events occuring at the site of application.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Guenthert, Prof. Dr. med., Principal Investigator
Locations (1):
- Dep. of Obstetrics and Gynecology, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Result] Gunthert AR, Limacher A, Beltraminelli H, Krause E, Mueller MD, Trelle S, Bobos P, Juni P. Efficacy of topical progesterone versus topical clobetasol propionate in patients with vulvar Lichen sclerosus - A double-blind randomized phase II pilot study. Eur J Obstet Gynecol Reprod Biol. 2022 May;272:88-95. doi: 10.1016/j.ejogrb.2022.03.020. Epub 2022 Mar 10. PMID 35290878